CLINICAL TRIAL: NCT01207206
Title: Oral Ketamine as an Adjuvant to Opioids for Pain Treatment in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Silviu Brill MD, Tel aviv Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-10-SB-392-CTIL
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2010-09

CONDITIONS: Cancer; Pain; Tolerance
Keywords: Patient suffering from severe cancer pain despite the opioid treatment; Opiate tolerance suspected on the basis of rapid escalation in opiate dose; Severe opiate side effects
MeSH Terms: conditions — Neoplasms; Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oral ketamine — The group will be divided into two pain matched groups of 25 each. One group will receive Ketamine (K group) and the other placebo (P). Both the researchers and the patients will not know to which group they belong. Four days prior to the beginning of the research the patients will document, using an ad-hoc diary, in predetermined hours, four times a day the level (VAS) of pain, sedation and vomiting scores, and other side effects. Pain will be assessed using a Visual Analog Scale (VAS) (0-10).
  The documentation will continue throughout the research period. The Ketamine or plaecebo will also be taken in a predetermined hours to avoid an effect of diurnal disruption on pain perception

SUMMARY:
In the current research the investigators would like to examine the effect of a well acquainted drug, Ketamine, which is used by anesthesiologists to induce sleep in operations. Usually the ketamine is given into the vein and not orally. The investigators want to give it orally to cancer patients that sufffer from severe pain to find out whether it can prove their quality of life, lower their pain and reduce the amount of opioids they receive.

DETAILED DESCRIPTION:
It is estimated that 10%-15% of patients with cancer-related pain do not achieve acceptable levels of pain relief even when oral or parenteral opioids are skillfully combined with conventional adjuvant analgesics and intractable pain occurs in up to 2% of advanced cancer patients. Painful conditions arising from tumor-nerve structure involvement, neuropathic pain, skin lesions, iatrogenic (chemo-and radiotherapy lesion), or ischemic pain are those most likely to require more aggressive treatment, such as the use of unconventional agents or interventional management approaches.

Despite considerable progress in the technologies of cancer-related pain management and an increased broadening array of medications, many patients fail to achieve adequate pain relief. In others, the availability of these treatments may be limited by such factors as side effects, or lack of or pain-management expertise. Furthermore, the development of opioid tolerance and the high incidence of side effects with escalating dose of opioid dose may contribute to treatment failure.

The need to develop new pharmacologic approaches for refractory pain remains of critical importance. The most potent class of analgesics available for general use remains the opioids.

Several lines of investigation have focused on the neuro-physiological as well as neuro-chemical mechanisms that may underlay opioid resistant pain, such as opioid induced hyperalgesia and opioid tolerance cause certain types of pain to be relatively resistant to the opioids or that may underlie the tolerance that can develop to their beneficial effects. Particular attention has been paid to the role played by glutamate neurotransmission in promoting and maintaining chronic pain states.

Glutamate is the primary excitatory neurotransmitter of the central nervous system and is normally released by pain-signaling afferent neurons as they synapse on central pain pathways in the spinal cord. The persistent release of glutamate, due to peripheral injury or inflammation, leads to the activation of N-methyl-D-aspartate (NMDA) receptors. This process of activation has been shown to play a crucial role in mediating the phenomenon of "wind up" pain, a state in which spinal neurons become hyper-responsive to repetitive painful stimulation.

The clinically observed phenomena of allodynia (pain due to a stimulus that does not normally provoke pain) and hyperalgesia (an increased response to a stimulus that is normally painful), which are the hallmarks of neuropathic pain, are expressions of "wind up" pain. Recent investigations indicate that this process can be prevented or mitigated by agents that block the effects of glutamate at the NMDA receptor. Other investigations have revealed that NMDA receptor antagonists can be useful in potentiating the analgesic efficacy of several classes of medication, including opioids, nonsteroidal anti-inflammatory drugs (NSAIDs), and local anesthetics. In addition, NMDA receptor antagonists may play an important role in mediating the development of opioid tolerance or in treating the perplexing syndrome of opiate-induced hyperalgesia.

Of the small number of NMDA receptor antagonists currently available for clinical use, most, unfortunately, either have a narrow therapeutic window or require parenteral administration. Dextromethorphan, best known for its use as an antitussive agent, is dosed orally and shows activity as a noncompetitive NMDA antagonist. Multiple trials, however, generally have not shown dextromethorphan to be effective in treating neuropathic pain.

Ketamine, a phencyclidine (PCP) derivative analog, has been used for more than 40 years to produce "dissociative" anesthesia.

Early experience with ketamine revealed that it also produced analgesia that sometimes well outlasted its anesthetic effects. Although the mechanisms of ketamine's analgesic effects remain the subject of debate, and are likely multiple, antagonism at the NMDA-receptor site appears to be central to both its anesthetic and analgesic effects.

Ketamine's utility as an anesthetic has been hampered by troublesome psychomimetic effects, which for many years have also limited its application as an analgesic. Recent investigations have shown, however, that analgesia can be produced with sub-hypnotic sub-anesthetic doses of intravenous ketamine (ie,10%-20% of those used for anesthesia) with a far lower frequency of psychomimetic reactions. These side effects are dose dependent and can be minimized by starting ketamine at low doses, titrating slowly, and concurrently starting a benzodiazepine or haloperidol.

Over the years a variety of nociceptive (somatic and visceral) and neuropathic pain states have been treated with subanesthetic doses of ketamine. Early studies demonstrated its utility in treating the pain associated with wound dressings in burn patients, as a treatment for pain following severe trauma and for cancer-related pain.

Racemic ketamine has an oral bioavailability of approximately 17%. When administrated orally in a dose of 0.5mg/kg the plasma ketamine concentration of ketamine was 40 ngml-1 (for the same i.m. dose the plasma ketamine concentration was 150 ng ml-1 ). Oral administration is associated with much greater concentrations of the metabolite norketamine, which may have contributed to the analgesic effect. Orally administered ketamine undergoes extensive first pass metabolism, primarily via N-de-methylation, resulting in low ketamine concentrations and high norketamine concentrations in blood and tissue. The plasma levels at which analgesia is achieved are 0.15 μg/ml following intramuscular administration and 0.04 μg/ml after oral administration. This difference may be explained by a higher norketamine concentration due to first-pass metabolism. This main metabolite apparently contributes to the antinociceptive effect Oral ketamine is more potent (30 to 40%) that subcutaneous route because first pass metabolism converts ketamine to an active analgesic metabolite.

The benefits and harms of adding ketamine to a strong analgesics pain-killers such as morphine for the relief of cancer pain are not yet established. Only two small randomised controlled trials suggest that when ketamine is given with morphine it may help to control cancer pain. However, these data are insufficient to assess the effectiveness of ketamine in this setting. So far there is little clinical evidence to support this practice, furthermore, the The Cochrane Database of Systematic Reviews 2009 concludes that: "Current evidence is insufficient to assess the benefits and harms of ketamine as an adjuvant to opioids for the relief of cancer pain. More randomized randomised controlled trials are needed".

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient suffering from severe cancer pain (VAS>6 at rest or on movement) despite the opioid treatment.

  2. Opiate tolerance suspected on the basis of rapid escalation in opiate dose 3. Severe opiate side effects

Exclusion Criteria:

* 1. Recent psychiatric hospitalization, suicide attempt, or history within the preceding month of electroconvulsive therapy 2. History of psychosis, eg, schizophrenia 3. History of recent seizures 4. Uncontrolled intracranial hypertension due to brain metastasis or hydrocephalus 5. Severe labile hypertension or poorly controlled cardiac arrhythmia 6. Chronic obstructive pulmonary disease (COPD) associated with hypercarbia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The capability of oral ketamine treatment to reduce pain | 4 months
  The study is a prospective randomized, placebo-controlled double -blind study involving. Subjects Fifty patients with unbalanced (VAS>6) chronic cancer-related pain despite opioid treatment.

SECONDARY OUTCOMES:
evaluation of side effects related to ketamine in cancer pain patients | 4 months
  The study is a prospective randomized, placebo-controlled double -blind study involving. Subjects Fifty patients with unbalanced (VAS>6) chronic cancer-related pain despite opioid treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel